CLINICAL TRIAL: NCT06232590
Title: Performance Comparison of Two Monthly Replacement Silicone Hydrogel Multifocal Lens Types
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision International Limited (CVIL) (Industry)
Collaborators: Centre for Ocular Research & Education, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-153
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-11

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Lens, then Test Lens (Experimental): Participants wore Control Lens for 1 month, then the Test Lens for 1 month
  Interventions: Device: Control Lens (comfilcon A); Device: Test Lens (lehfilcon A)
- Test Lens, then Control Lens (Experimental): Participants wore the Test Lens for 1 month, then the Control Lens for 1 month
  Interventions: Device: Control Lens (comfilcon A); Device: Test Lens (lehfilcon A)

INTERVENTIONS:
Device: Control Lens (comfilcon A) — Multifocal monthly replacement contact lens for 1 month
Device: Test Lens (lehfilcon A) — Multifocal monthly replacement contact lens for 1 month

SUMMARY:
To evaluate and compare the performance of two monthly replacement multifocal contact lenses in existing wearers.

DETAILED DESCRIPTION:
This was a prospective, randomized, participant-masked, crossover, bilateral dispensing study. Each lens type was worn for approximately 4-6 weeks: the lens prescription of each lens type was optimized after 3-10 days wearing experience, prior to starting a 1-month (28-32 days) wear period.

ELIGIBILITY:
Inclusion Criteria:

1. Were at least 42 years of age and had full legal capacity to volunteer;
2. Had read and signed an information consent letter;
3. Self-reported having had a full eye examination in the previous two years;
4. Anticipated being able to wear the study lenses for at least 8 hours a day, 5 days a week;
5. Were willing and able to follow instructions and maintain the appointment schedule;
6. Habitually wore spherical multifocal soft contact lenses, for the past 3 months minimum:

   * Maximum of 4 participants (out of 12) per site could be habitual wearers of daily disposable lenses,
   * Maximum of 4 participants (out of 12) per site could be habitual wearers of Biofinity Multifocal,
   * Maximum of 4 participants (out of 12) per site could be habitual wearers of either TOTAL30 Multifocal or AirOptix plus HydraGlyde Multifocal
7. Had refractive astigmatism no higher than -0.75DC;
8. Is presbyopic and requires a reading addition of at least +0.75D and no more than +2.50D;
9. Could be fit and achieve binocular distance vision of at least 20/30 Snellen which participants also deem to be 'acceptable', with the available study lens parameters (Distance sphere +4 to -6; near addition as per study design).

Exclusion Criteria:

1. Were participating in any concurrent clinical or research study;
2. Had any known active ocular disease and/or infection that contraindicated contact lens wear;
3. Had a systemic or ocular condition that in the opinion of the investigator may have affected a study outcome variable;
4. Were using any systemic or topical medications that in the opinion of the investigator may have affect contact lens wear or a study outcome variable;
5. Had known sensitivity to the diagnostic sodium fluorescein used in the study;
6. Self-reported as pregnant, lactating or planning a pregnancy at the time of enrolment;
7. Had undergone refractive error surgery or intraocular surgery.

Min Age: 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sacco, Principal Investigator — Sacco Eye Group; David Wilkinson, Principal Investigator — Spadina Optometry; Katherine Bickle, Principal Investigator — ProCare Vision Center; Dustin Gardner, Principal Investigator — New Bremen EyeCare; Gina Wesley, Principal Investigator — Complete Eye Care of Medina
Locations (5):
- United States (4):
  - Complete Eye Care of Medina, Medina, Minnesota
  - Sacco Eye Group, Vestal, New York
  - ProCare Vision Center, Granville, Ohio
  - New Bremen EyeCare, New Bremen, Ohio
- Spadina Optometry, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Lens, Then Test Lens: Participants wore the Control Lens for 1 month, then the Test Lens for 1 month
Period: Period 1: First Intervention
Arm/Group | Control Lens, Then Test Lens | Test Lens, Then Control Lens
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0
Period: Period 2: Second Intervention
Arm/Group | Control Lens, Then Test Lens | Test Lens, Then Control Lens
Started | 30 | 30
Completed | 29 | 30
Not Completed | 1 | 0
Not completed — Unable to attend study visit | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Participants who completed all study visits.
Arm/Group | Overall Study
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Lens Handling for Insertion
Description: Subjective rating collected in office using a 0-100 scale, where 0=Very difficult and 100=Very easy. The participant rated the study lens considering a typical day in the last 1 month of wear.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Lens: Participants that received the Control Lens and completed all study visits.
- Test Lens: Participants that received the Test Lens and completed all study visits.
Arm/Group | Control Lens | Test Lens
Number analyzed (Participants) | 59 | 59
score on a scale | 95 (9) | 96 (8)

ADVERSE EVENTS:
Time Frame: Length of study, approximately 3 months
Groups:
- Control Lens: All participants that received the Control Lens.
- Test Lens: All participants that received the Test Lens.
Arm/Group | Control Lens | Test Lens
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/59
Other Adverse Events (participants affected / at risk) | 4/60 | 4/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Lens (N=60) | Test Lens (N=59)
Small lymph cysts (Eye disorders) | 0 (0) | 1 (2)
Subconjunctival hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Eye floaters (Eye disorders) | 0 (0) | 1 (1)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Stomach distress (Gastrointestinal disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Primary care provider intervention (Surgical and medical procedures) | 1 (1) | 0 (0) — Per primary care providers recommendation participant stopped the medication Vyvanse.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/90/NCT06232590/Prot_SAP_000.pdf